CLINICAL TRIAL: NCT01565928
Title: A PHASE 1B, OPEN-LABEL, SAFETY AND TOLERABILITY STUDY OF ORAL MDV3100 IN COMBINATION WITH DOCETAXEL IN MEN WITH ADVANCED PROSTATE CANCER
Brief Title: Safety and Tolerability Study of MDV3100 in Combination With Docetaxel in Men With Advanced Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry); Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDV3100-06; C3431002 (Other: Alias Study Number)
Record Dates: First submitted 2012-02-08; First posted 2012-03-29 (Estimated); Results first posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; docetaxel; MDV3100; enzalutamide; Xtandi
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MDV3100 (Experimental)
  Interventions: Drug: MDV3100

INTERVENTIONS:
Drug: MDV3100 — 4 x 40 mg capsules, orally, once per day

SUMMARY:
The purpose of this study is to determine the safety of MDV3100 given in combination with Docetaxel in men with advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent;
* Men, 18 years of age or older;
* Histologically or cytologically confirmed adenocarcinoma of the prostate;
* Ongoing androgen deprivation therapy

Exclusion Criteria:

* Severe concurrent disease;
* Known or suspected brain metastasis;
* History of another malignancy within the previous 5 years;
* Prior treatment with docetaxel-based chemotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 23 (Actual)
Dates: Start 2012-01-24 (Actual); Primary Completion 2013-07-01 (Actual); Study Completion 2018-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Virginia Oncology Associates, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel 75 mg/m^2+ Enzalutamide 160 mg: Docetaxel 75 milligrams per square meter (mg/m^2) was administered as intravenous (IV) infusion for 1 hour on Day 1 of each treatment period (each treatment period was of 21 days). From Day 2 of treatment period 1, participants received a single oral dose of Enzalutamide (MDV3100) 160 milligrams (mg) (4 capsules of 40 mg each) once daily. Participants received a single oral dose of Dexamethasone 8 mg prior to each Docetaxel infusion and Prednisone (5 mg) once daily on the days of Docetaxel administration then twice daily every day thereafter as long as Docetaxel treatment continued. Participants who tolerated treatment with Docetaxel and Enzalutamide continued to receive the combined therapy. Participants who discontinued Docetaxel were allowed to continue the treatment with Enzalutamide 160 mg once daily up to the end of study treatment (maximum of Month 70).
Period: Overall Study
Arm/Group | Docetaxel 75 mg/m^2+ Enzalutamide 160 mg
Started | 22
Completed | 0
Not Completed | 22
Not completed — Adverse Event | 3
Not completed — Other | 3
Not completed — Progressive Disease | 13
Not completed — Withdrawal by Subject | 1
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all enrolled participants.
Arm/Group | Docetaxel 75 mg/m^2+ Enzalutamide 160 mg
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (10.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Required Study Drug Dose Reduction During Treatment Periods 1 and 2
Description: Percentage of participants that required dose reductions of Docetaxel and Enzalutamide treatment were reported in this outcome measure. Dose modifications (interruptions or dose reductions) were permitted for participants who had adverse events that were intolerable or could not be improved by other means. Dose reductions or delays were determined according to the prescribing information and at the discretion of the investigator.
Time Frame: Treatment Period 1 (Day 1) up to end of Treatment Period 2 (42 days)
Population: Safety population included all enrolled participants who received at least 1 dose or partial dose of study drug (Enzalutamide and/or Docetaxel).
Measure: Number; unit: percentage of participants
Groups:
- Combination Therapy: Docetaxel 75 mg/m^2+ Enzalutamide 160 mg: Docetaxel 75 mg/m^2 was administered as IV infusion for 1 hour on Day 1 in each treatment period (each treatment period was of 21 days). From Day 2 of treatment Period 1 participants received a single oral dose of Enzalutamide 160 mg once daily. Participants received a single oral dose of Dexamethasone 8 mg prior to each Docetaxel infusion and Prednisone 5 mg once daily on the days of docetaxel administration then twice daily every day thereafter as long as docetaxel treatment continued. Participants who tolerated treatment with Docetaxel and Enzalutamide received the both.
Arm/Group | Combination Therapy: Docetaxel 75 mg/m^2+ Enzalutamide 160 mg
Number analyzed (Participants) | 22
percentage of participants
  Docetaxel Dose Reductions | 4.5
  Enzalutamide Dose Reductions | 0.0

2. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event (AE)
Description: AE was any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Percentage of participants that discontinued study drug due to adverse events were reported in this outcome measure.
Time Frame: Treatment Period 1 (Day 1) up to end of study treatment (maximum 70 months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel 75 mg/m^2+ Enzalutamide 160 mg
Number analyzed (Participants) | 22
percentage of participants | 9.1

3. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Criteria:1)systolic blood pressure (SBP):a) absolute result(AR)>=180millimeters of mercury(mmHg) and increase from baseline(BL)greater than(>)40mmHg,b)less than(<)90mmHg and decrease from BL>30mmHg,c)most extreme post-BL result>=140mmHg,d)most extreme post-BL result>=180mmHg,e)most extreme result(MER)>=180mmHg and >=20mmHg change from BL,f)MER>=140mmHg and >=20mmHg change from BL;2)diastolic blood pressure(DBP):a)AR>105mmHg and increase from BL,b)AR<50mmHg and decrease from BL>20mmHg;c)most extreme post-BL result>=90mmHg,d)MER>=90mmHg and >=15mmHg change from BL,e)most extreme post-BL result>=105mmHg,f)MER>=105mmHg and>=15mmHg change from BL;3)heart rate:a)AR>120 beats per minute(bpm) and increase from BL>30bpm,b) AR<50 bpm and decrease from BL>20bpm.Only those categories in which at least 1 participant had clinically significant vital sign abnormality, were reported in this outcome measure.T1 = Timeframe for "Combination Therapy" and T2 = Time frame for "Post-Docetaxel Enzalutamide".
Time Frame: T1= Baseline (Day 1) up to a maximum of approximately Month 12; T2 = From Month 10.6 up to a maximum of approximately Month 71.5
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Post-Docetaxel Enzalutamide 160 mg: Participants who had received the combination therapy of Docetaxel and Enzalutamide but discontinued the Docetaxel treatment and continued to receive a single oral dose of Enzalutamide 160 mg (4 capsule each of 40 mg) once daily up to the end of the study treatment (maximum of 70 months).
Arm/Group | Combination Therapy: Docetaxel 75 mg/m^2+ Enzalutamide 160 mg | Post-Docetaxel Enzalutamide 160 mg
Number analyzed (Participants) | 22 | 21
Participants
  SBP: AR- > 180 mmHg, increase from BL > 40 mmHg | 0 | 1
  SBP: AR- < 90 mmHg, decrease from BL > 30 mmHg | 1 | 0
  SBP: Most extreme post- BL result >= 140 mmHg | 10 | 7
  SBP: Most extreme post- BL result >= 180 mmHg | 0 | 2
  SBP: MER >= 180 mmHg, >= 20 mmHg change from BL | 0 | 2
  SBP: MER >= 140 mmHg, >= 20 mmHg change from BL | 5 | 5
  DBP: Most extreme post-BL result >= 90 mmHg | 3 | 6
  DBP: Most extreme post-BL result >= 105 mmHg | 0 | 1
  DBP: MER >= 105 mmHg,>= 15 mmHg change from BL | 0 | 1
  DBP: MER >= 90 mmHg,>= 15 mmHg change from BL | 1 | 4
  Heart Rate: AR >120 bpm, increase from BL >30 bpm | 0 | 1
  Heart Rate: AR <50 bpm, decrease from BL >30 bpm | 0 | 1

4. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Electrocardiograms (ECG)
Description: Clinically significant changes from baseline in ECG findings was based up on investigator's discretion. T1 = Timeframe for "Combination Therapy: Docetaxel 75 mg/m^2+ Enzalutamide 160 mg" and T2 = Time frame for "Post-Docetaxel Enzalutamide 160 mg".
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy: Docetaxel 75 mg/m^2+ Enzalutamide 160 mg | Post-Docetaxel Enzalutamide 160 mg
Number analyzed (Participants) | 22 | 21
Participants | 1 | 0

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Docetaxel With and Without Enzalutamide Treatment
Time Frame: Docetaxel without Enzalutamide: Predose, 0.5, 1, 1.5, 2, 4, 8 and 24 hour post docetaxel infusion on Day 1 of Treatment Period 1; Docetaxel with Enzalutamide: Predose, 0.5, 1, 1.5, 2, 4, 8 and 24 hour post docetaxel infusion on Day 1 of Treatment Period 2
Population: Pharmacokinetic (PK) population included all enrolled participants who received at least 2 doses of Docetaxel (75 mg/m^2) and underwent PK sampling after both doses. Here, 'Number analyzed' signifies number of participants who were evaluable for the specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Combination Therapy: Docetaxel 75 mg/m^2+ Enzalutamide 160 mg
Number analyzed (Participants) | 22
nanograms per milliliter
  Docetaxel Without Enzalutamide | 1722.1 (27.14)
  Docetaxel With Enzalutamide: number analyzed (Participants) | 18
  Docetaxel With Enzalutamide | 1662.9 (23.00)

6. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUClast) of Docetaxel With and Without Enzalutamide Treatment
Description: AUClast was observed using a linear mixed-effects model.
Time Frame: as for outcome 5
Population: PK population included all enrolled participants who received at least 2 doses of Docetaxel (75 mg/m^2) and underwent PK sampling after both doses. Here, 'Number analyzed' signifies number of participants who were evaluable for the specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter
Arm/Group | Combination Therapy: Docetaxel 75 mg/m^2+ Enzalutamide 160 mg
Number analyzed (Participants) | 22
nanograms*hour per milliliter
  Docetaxel Without Enzalutamide | 1866.6 (29.05)
  Docetaxel With Enzalutamide: number analyzed (Participants) | 18
  Docetaxel With Enzalutamide | 1674.4 (19.32)

7. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinite Time (AUCinf) of Docetaxel With and Without Enzalutamide Treatment
Description: AUCinf was observed using a linear mixed-effects model.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter
Arm/Group | Combination Therapy: Docetaxel 75 mg/m^2+ Enzalutamide 160 mg
Number analyzed (Participants) | 22
nanograms*hour per milliliter
  Docetaxel Without Enzalutamide | 2020.1 (27.98)
  Docetaxel With Enzalutamide: number analyzed (Participants) | 18
  Docetaxel With Enzalutamide | 1769.1 (18.91)

ADVERSE EVENTS:
Time Frame: Baseline up to a maximum of approximately Month 12 for Combination Therapy; From Month 10.6 up to a maximum of approximately Month 71.5 for Post-Docetaxel Enzalutamide
Description: An event may be categorized as serious in one participant and non-serious in another, or 1 participant may experience both event. All treatment emergent AEs and SAEs were collected and reported. The same event may appear as both AE and SAE. Safety population included all enrolled participants who received at least 1 dose or partial dose of study drug (Enzalutamide and/or Docetaxel).
Arm/Group | Combination Therapy: Docetaxel 75 mg/m^2+ Enzalutamide 160 mg | Post-Docetaxel Enzalutamide 160 mg
Serious Adverse Events (participants affected / at risk) | 8/22 | 7/21
Other Adverse Events (participants affected / at risk) | 21/22 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy: Docetaxel 75 mg/m^2+ Enzalutamide 160 mg (N=22) | Post-Docetaxel Enzalutamide 160 mg (N=21)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 2 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 3
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
ASTHENIA (General disorders) | 0 | 1
DEATH (General disorders) | 1 | 0
IMPAIRED HEALING (General disorders) | 0 | 1
PYREXIA (General disorders) | 1 | 1
CELLULITIS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 1
SEPSIS (Infections and infestations) | 1 | 1
SEPTIC SHOCK (Infections and infestations) | 0 | 1
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 1 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 1
OBSTRUCTIVE UROPATHY (Renal and urinary disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 0
ARTERIOSCLEROSIS (Vascular disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy: Docetaxel 75 mg/m^2+ Enzalutamide 160 mg (N=22) | Post-Docetaxel Enzalutamide 160 mg (N=21)
ANAEMIA (Blood and lymphatic system disorders) | 4 | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 19 | 1
CATARACT (Eye disorders) | 0 | 2
LACRIMATION INCREASED (Eye disorders) | 5 | 2
VISION BLURRED (Eye disorders) | 2 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 3
CONSTIPATION (Gastrointestinal disorders) | 7 | 9
DIARRHOEA (Gastrointestinal disorders) | 6 | 0
DYSPEPSIA (Gastrointestinal disorders) | 4 | 1
NAUSEA (Gastrointestinal disorders) | 9 | 1
STOMATITIS (Gastrointestinal disorders) | 3 | 0
ASTHENIA (General disorders) | 3 | 1
CHEST PAIN (General disorders) | 2 | 1
FATIGUE (General disorders) | 16 | 5
INFLUENZA LIKE ILLNESS (General disorders) | 2 | 0
OEDEMA (General disorders) | 2 | 2
OEDEMA PERIPHERAL (General disorders) | 3 | 2
PAIN (General disorders) | 4 | 1
PYREXIA (General disorders) | 1 | 2
CELLULITIS (Infections and infestations) | 1 | 1
OSTEOMYELITIS (Infections and infestations) | 0 | 2
RHINITIS (Infections and infestations) | 1 | 1
URINARY TRACT INFECTION (Infections and infestations) | 2 | 0
BLOOD CREATININE INCREASED (Investigations) | 1 | 1
BLOOD PHOSPHORUS DECREASED (Investigations) | 2 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 3 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 5 | 6
DEHYDRATION (Metabolism and nutrition disorders) | 3 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 2
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 | 5
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 2
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 3 | 2
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 2 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 | 5
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 3
DIZZINESS (Nervous system disorders) | 4 | 1
DYSGEUSIA (Nervous system disorders) | 6 | 1
HEADACHE (Nervous system disorders) | 3 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 10 | 1
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 3 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 7 | 4
DEPRESSION (Psychiatric disorders) | 0 | 2
INSOMNIA (Psychiatric disorders) | 4 | 1
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 2 | 2
INCONTINENCE (Renal and urinary disorders) | 1 | 1
POLLAKIURIA (Renal and urinary disorders) | 3 | 3
URETHRAL PAIN (Renal and urinary disorders) | 0 | 2
PELVIC PAIN (Reproductive system and breast disorders) | 0 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 | 4
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 4 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 6 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 1
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 3 | 1
RASH (Skin and subcutaneous tissue disorders) | 3 | 3
HOT FLUSH (Vascular disorders) | 1 | 2
HYPERTENSION (Vascular disorders) | 1 | 1
HYPOTENSION (Vascular disorders) | 1 | 1
INTERMITTENT CLAUDICATION (Vascular disorders) | 2 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
DEAFNESS (Ear and labyrinth disorders) | 1 | 0
TINNITUS (Ear and labyrinth disorders) | 0 | 1
BLEPHAROSPASM (Eye disorders) | 1 | 0
DRY EYE (Eye disorders) | 1 | 0
EYE IRRITATION (Eye disorders) | 1 | 0
EYE PRURITUS (Eye disorders) | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1
FAECES DISCOLOURED (Gastrointestinal disorders) | 1 | 0
FLATULENCE (Gastrointestinal disorders) | 1 | 0
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 | 1
OESOPHAGEAL PAIN (Gastrointestinal disorders) | 1 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 1
ORAL DISORDER (Gastrointestinal disorders) | 0 | 1
PARAESTHESIA ORAL (Gastrointestinal disorders) | 1 | 0
CATHETER SITE ERYTHEMA (General disorders) | 1 | 0
CHILLS (General disorders) | 1 | 0
GAIT DISTURBANCE (General disorders) | 1 | 0
GENERALISED OEDEMA (General disorders) | 0 | 1
IMPAIRED HEALING (General disorders) | 1 | 0
MEDICAL DEVICE PAIN (General disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 0
FURUNCLE (Infections and infestations) | 1 | 0
HEPATOSPLENIC CANDIDIASIS (Infections and infestations) | 0 | 1
INFUSION SITE INFECTION (Infections and infestations) | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 0 | 1
MUCOSAL INFECTION (Infections and infestations) | 0 | 1
ORAL INFECTION (Infections and infestations) | 0 | 1
SKIN INFECTION (Infections and infestations) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 1
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 1
BLOOD CALCIUM DECREASED (Investigations) | 1 | 0
BLOOD CHOLESTEROL INCREASED (Investigations) | 0 | 1
BLOOD GLUCOSE DECREASED (Investigations) | 1 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 1
BLOOD MAGNESIUM DECREASED (Investigations) | 1 | 0
BLOOD POTASSIUM INCREASED (Investigations) | 1 | 1
BLOOD URIC ACID INCREASED (Investigations) | 1 | 0
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1 | 0
WEIGHT DECREASED (Investigations) | 1 | 0
ACIDOSIS (Metabolism and nutrition disorders) | 0 | 1
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 1
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 0 | 1
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 | 0
AMNESIA (Nervous system disorders) | 1 | 0
APHASIA (Nervous system disorders) | 0 | 1
BALANCE DISORDER (Nervous system disorders) | 1 | 0
COGNITIVE DISORDER (Nervous system disorders) | 0 | 1
HYPOKINESIA (Nervous system disorders) | 0 | 1
PARAESTHESIA (Nervous system disorders) | 0 | 1
AGITATION (Psychiatric disorders) | 0 | 1
BLADDER SPASM (Renal and urinary disorders) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 1
NIPPLE DISORDER (Reproductive system and breast disorders) | 0 | 1
SCROTAL OEDEMA (Reproductive system and breast disorders) | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 1
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1 | 0
ONYCHOMADESIS (Skin and subcutaneous tissue disorders) | 1 | 0
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 1
ARTERIOSCLEROSIS (Vascular disorders) | 0 | 1
FLUSHING (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.